CLINICAL TRIAL: NCT02749565
Title: he Role of Endothelium A and EGFR Receptor in Fibrocytes From Asthma With Obstructive Sleep Apnea
Brief Title: The Role of Endothelium A and EGFR Receptor in Fibrocytes From Asthma With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 102-5744A3
Record Dates: First submitted 2016-04-07; First posted 2016-04-25 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-11

CONDITIONS: Asthma; OSA
Keywords: asthma; fibrocyte; airway remodeling; OSA; hypoxia
MeSH Terms: conditions — Asthma; Airway Remodeling; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — circulating fibrocytes purified from PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- asthmatic patients with OSA
- asthmatic patients without OSA

SUMMARY:
The investigators will compare the circulating fibrocyte proportion in asthmatic patients with obstructive sleep apnea (OSA) and not with OSA In addition, the investigators will compare the expression of epidermal growth factor receptor (EGFR), endothelin A receptor (ETAR) and connective tissue growth factor (CTGF) The association of those factors and annual decline of forced expiratory volume in 1 second (FEV1) will be performed

DETAILED DESCRIPTION:
Asthma is characterized by airflow obstruction, chronic airway inflammation and remodeling. The investigators' report has shown directly the relationship between fibrocytes, and chronic airflow obstruction with rapid decline in FEV1 in asthma. Asthma concomitant of obstructive sleep apnea (OSA) may appear intermittent hypoxia and result in the frequent attack of asthma symptoms. In animal model, hypoxia may increase the circulating fibrocytes, thus play a role in pulmonary hypertension. The investigators' published paper also showed that an increased expression of EGFR, ETAR and Vascular endothelial growth factor receptor (VEGFR) in circulating fibrocytes in chronic obstructive asthmatics. It is unknown whether circulating fibrocytes from asthma with OSA have the higher expression of EGFR, connective tissue growth factor receptor, VEGFR and ETAR compared to asthma without OSA. The investigators are also interested in whether proliferation and differentiation of fibrocytes are different between asthmatics with or without concomitant of OSA. The investigators will study the correlation between the percentage of circulating fibrocytes and the oxygen desaturation index (ODI) and severity of sleep apnea to clarify the role of hypoxia, which contributing to chronic asthma.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of asthma

Exclusion Criteria:

* chronic obstructive pulmonary disease (COPD)
* bronchiectasis
* cystic fibrosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the diagnosis of asthma based on current or past smoking history, clinical evaluation, and pulmonary function testing showing airflow obstruction (FEV1/FVC < 70%) with a change in FEV1 of large than 200 ml and 12% in the bronchodilator test will be enrolled.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
circulating fibrocyte proportion between asthmatic patient with OSA and without OSA | baseline

SECONDARY OUTCOMES:
the change of circulating fibrocyte proportion in asthmatic patients with OSA | baseline

CONTACTS AND LOCATIONS:
Overall Officials: TSAI-YU WANG, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No